CLINICAL TRIAL: NCT06292273
Title: Bupivacaine With Dexmedetomidine Versus Bupivacaine Alone for Transversus Abdominis Plane Block for Post-operative Analgesia in Patients Undergoing Caesarean Section: A Comparative Study.
Brief Title: Bupivacaine With Dexmedetomidine Versus Bupivacaine Alone for Transversus Abdominis Plane Block in Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, rabab Mohammad habeeb, Principal investigator, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ANET19
Record Dates: First submitted 2024-02-21; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: randomized, double blind case control
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Bupivacain Plus dexamethasone (Active Comparator): receiving plain bupivacaine 0.1%, 35 ml with dexmedetomidine 0.5
  Interventions: Procedure: Transversus Abdominis Plane Block with bupivacain Plus dexamethasone
- Group bupivacain (Placebo Comparator): plain bupivacaine 0.25%, 25 ml bilaterally
  Interventions: Procedure: Transversus Abdominis Plane Block with bupivacain

INTERVENTIONS:
Procedure: Transversus Abdominis Plane Block with bupivacain Plus dexamethasone — Bupivacain 0.1%, 35 ml with dexmedetomidine 0.5 µG/kg on each side
  Arms: Group Bupivacain Plus dexamethasone
Procedure: Transversus Abdominis Plane Block with bupivacain — plain bupivacaine 0.25%, 25 ml bilaterally
  Arms: Group bupivacain

SUMMARY:
Transversus Abdominis plane (TAP) block is a regional technique for providing analgesia of the anterolateral abdominal wall. TAP block are commonly given in patients who have undergone various abdominal as well as pelvic surgeries such as caesarean section, hysterectomy, appendicectomy and various laparoscopic surgeries. this study is conducted to analyse the effect of addition of dexmedetomidine to bupivacaine in Transversus Abdominis Plane (TAP) block.

DETAILED DESCRIPTION:
Peripheral nerve block is becoming increasingly popular technique for postoperative pain relief and is also established as a part of multimodal analgesia and enhanced recovery program. Transversus abdominis plane (TAP) block is a regional technique for providing analgesia of the anterolateral abdominal wall. TAP block are commonly given in patients who have undergone various abdominal as well as pelvic surgeries such as caesarean section, hysterectomy, appendicectomy and various laparoscopic surgeries.The Purpose of a TAP block is to infiltrate local anaesthetic agents in the plane between the internal oblique and transversus abdominis muscles thereby providing effective postoperative analgesia. Earlier the blind TAP block (through lumbar triangle of Petit) was commonly given but with widespread use of ultrasound nowadays it is almost always given under ultrasound guidance. Accuracy and efficacy of TAP block is significantly improved under ultrasound guidance because under ultrasound guidance the anesthetic agent can be properly deposited in the neurovascular plane. Ultrasound provides real time and direct visualisation of needle during infiltration of local anaesthetic drug.

ELIGIBILITY:
Inclusion Criteria:

* pregnant female elected for cesarean section
* ASAll

Exclusion Criteria:

* coagulopathy
* BMI>35

  * heart Diseases
  * diabets

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Post operative pain | 24 hours
  visual analog score from 0 to 10 where 0 is no pain and 10 worst pain ever

SECONDARY OUTCOMES:
Sedation | 24 hours
  Modefied Ramsey sedation score from 1 to 6
Heart rate | 24 hours
  pulse/ min
Total analgesic consumption | 24 hours
  Mg
Side effects | 24hours
  Nausea, vomiting, pruritus

CONTACTS AND LOCATIONS:
Overall Officials: rabab M habeeb, Principal Investigator — Menoufia University
Locations (1):
- Faculty of Medicine Menoufia University, Cairo, Governorate, Egypt